CLINICAL TRIAL: NCT01633723
Title: A Phase I, Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dosing, Dose Escalation Clinical Trial With Open-labelled Food Effect Study of Single Dose to Investigate the Safety, Tolerability and Pharmacokinetics of DA-6886 After Oral Administration in Healthy Male Subjects
Brief Title: Phase I Clinical Trial of DA-6886 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DA6886_IBS_I
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — N-((1-(3-(1,2,3-triazol-1-yl)propyl)piperidin-4-yl)methyl)-4-amino-5-chloro-2-methoxybenzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DA-6886 (Experimental)
  Interventions: Drug: DA-6886
- DA-6886 placebo (Placebo Comparator)
  Interventions: Drug: Placebo of DA-6886

INTERVENTIONS:
Drug: DA-6886 — single dose study : DA-6886 1mg,2.5mg,5mg,10mg,20mg dosage (Dose-escalation)
  multiple dose study : DA-6886 2.5mg,5mg,10mg or 5mg,10mg,20mg dosage (Dose-escalation)
  Arms: DA-6886
Drug: Placebo of DA-6886 — DA-6886 placebo
  Arms: DA-6886 placebo

SUMMARY:
DA-6886_IBS_I is a phase I, dose block-randomized, double-blind, placebo-controlled, single/multiple dosing, dose escalation clinical trial with open-labelled food effect study of single dose to investigate the safety, tolerability and pharmacokinetics of DA-6886 after oral administration in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* 20 ~ 45 years old
* 27kg/m2 ≥ BMI ≥ 20kg/m2
* Healthy Male
* Informed consent

Exclusion Criteria:

* Clinically significant medical history
* smokers
* Clinically significant hypersensitivity of Drugs
* Clinically significant cutaneous disorder
* QTcB > 450msec
* have a history of drug abuse or show positive for drug abuse or cotinine at urine screening

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assessment of safety | up to 7 days (single dose study, single dose study for food effect), 15 days (multiple dose study)
  1. Adverse Events
  2. Laboratory Results
  3. Vital sign, Physical Examination, EKG

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | up to 48 hours after last dosing of DA-6886
  Cmax, Tmax, AUClast, Ae, Cssmax, Cssmin

CONTACTS AND LOCATIONS:
Locations (1):
- ASAN medical center, Seoul, Songpa-gu, South Korea